CLINICAL TRIAL: NCT01509313
Title: A Randomised Controlled Trial Comparing Morcellation With Electrical Resection for Removal of Uterine Polyps
Brief Title: A Trial Comparing Morcellation With Electrical Resection for Removal of Uterine Polyps
Acronym: MERT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Birmingham Women's NHS Foundation Trust (Other Government)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Thomas Justin Clark, Consultant Obstetrics and Gynaecologist, Birmingham Women's NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPS-MERT-01
Record Dates: First submitted 2012-01-05; First posted 2012-01-13 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Endometrial Polyps
Keywords: endometrial polyps; uterine polyps; morcellator; hysteroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uterine polypectomy using morcellator (Experimental): A new instrument using a mechanical cutting edge has come to market for uterine polypectomy. In patients having a general anaesthesia the mechanical cutting instrument has been shown to be easier to learn, more effective at completely removing polyps and quicker than current techniques. However, the instrument is slightly larger, which could potentially cause more discomfort and prolong the procedure in the outpatient setting.
  Interventions: Device: hysteroscopic morcellator (TruClear)
- Electical Resection (Active Comparator): At present the most commonly used device for removing the uterine polyps in the outpatient setting is by electrical resection. This will provide comparison for the morcellator device being tested
  Interventions: Device: Bipolar Electrical resectoscope (Versapoint)

INTERVENTIONS:
Device: hysteroscopic morcellator (TruClear) — It can be used to treat uterine pathology with a mechanical cutting edge
  Other Names: TruClear(Smith&Nephew, USA)
  Arms: Uterine polypectomy using morcellator
Device: Bipolar Electrical resectoscope (Versapoint) — It can be used to treat uterine pathology with an electrical cutting edge
  Other Names: Versapoint® (Gynecare; Ethicon Inc., New Jersey, USA).
  Arms: Electical Resection

SUMMARY:
Outpatient polyp treatment can be performed in a few different ways but generally involves passing a special type of hysteroscope (3-6 millimetre in diameter) into the womb through which specifically designed miniature operating instruments are passed to remove the polyp(s). At present the most commonly used instruments use an electrical cutting edge. However, a new instrument using a mechanical cutting edge has come to market. In patients having a general anaesthesia the mechanical cutting instrument has been shown to be easier to learn, more effective at completely removing polyps and quicker. However, the instrument is slightly larger, which could potentially cause more discomfort and prolong the procedure in the outpatient setting. Therefore, the investigators want to compare the electrical and mechanical instruments for speed, completeness of polyp removal and patient acceptability.

DETAILED DESCRIPTION:
The miniaturisation of hysteroscopes and ancillary instrumentation coupled with enhanced visualisation has enabled hysteroscopic surgery to be performed in an outpatient setting without the need for general anaesthesia or inpatient hospital admission. The most common operative hysteroscopic procedure is endometrial polypectomy and the feasibility and acceptability of such approaches has been demonstrated. The procedure involves removing polyps from the uterine cavity. Over 90% of UK gynaecologists routinely recommend removal of endometrial polyps following diagnosis with the aim of treating associated symptoms of abnormal bleeding and retrieving the specimen to exclude malignant or pre-malignant disease. The investigators have recently completed recruitment to a large, multicentre, randomised control trial called the Outpatient Polypectomy Trial ('OPT' http://www.opt.bham.ac.uk, ISRCTN65868569), which has compared treatment settings for the removal of endometrial polyps. Over 500 women were randomised between outpatient procedures and day-case procedures which require a general anaesthetic. The analysis regarding relative treatment effectiveness will be available in late 2012. Interestingly, this trial also recruited women who expressed a preference for treatment setting. This resulted in an additional 400 women entering the study of which over 90% had a preference for an outpatient setting (Personal communication Clark TJ).

Thus outpatient removal of polyps is, feasible, safe and preferred by women. The majority of gynaecologists performing outpatient procedures, cut polyps away from their attachment to the uterine wall using a miniature bipolar electrosurgical instrument; Versapoint® (Gynecare; Ethicon Inc., New Jersey, USA). This procedure is carried out under direct hysteroscopic vision, without the need for routine, potentially painful, dilatation of the cervix. Whilst the technology is feasible and effective it requires skill and experience in outpatient hysteroscopic surgery, which many UK gynaecologists lack and this is reflected in the limited adoption of outpatient procedures in spite of evidence supporting their use. Moreover, even for the experienced operator, retrieving the removed polyp specimen from the uterine cavity, to send off for histopathological assessment, can be a challenge due to the small operating field and the need to negotiate the narrower endocervical canal. Various methods are used to retrieve specimens and include the use of mechanical instruments (e.g. grasping forceps or snares) which do not require the cervix to be dilated. However, this approach often fails because of the fragility of these minute hysteroscopic instruments (diameter 1.2-1.8mm) so recourse to insertion of larger 'polyp' forceps blindly into the uterine cavity is necessary. The latter approach requires the use of local injection of anaesthetic into the cervix which is uncomfortable and dilatation of the cervix with the potential for uterine trauma.

Since, completion of recruitment of OPT trial a new technology has become available called the TRUCLEAR hysteroscopic morcellator (Smith&Nephew, Andover MASS, USA). This technology incorporates a 4mm disposable mechanical cutting device which simultaneously cuts and aspirates polyp tissue. The ability to both cut and retrieve polyps avoids the need for additional instrumentation of the uterine cavity in order to retrieve the detached polyp specimen i.e. a single insertion of the hysteroscope is required only. The use of mechanical morcellation may also improve visualisation during surgery by avoidance of bubble formation or the production of tissue fragments ('chips') associated with the electrosurgical approach. Thus, this new technology has potential advantages for the patient (acceptability, pain, infection, safety), the surgeon (speed, feasibility, completeness of the procedure) and health service (avoidance of second stage procedures under general anaesthetic). However, the established single use bipolar electrode is smaller than the disposable morcellator cutting device (1.6mm vs. 2.9mm). Moreover, the bipolar electrode can be used down the operating channel of a variety of continuous flow hysteroscopes which are longer and smaller in diameter and in day-to-day use in gynaecological practice in outpatient settings (outer diameter 4.1mm (Gynecare; Ethicon Inc., New Jersey, USA), 5mm Storz Bettocci hysteroscope (Karl Storz Endoscopy-America inc., California, USA) or Olympus 5.5mm (Olympus Corporation, Shinjuku-ku, Tokyo, Japan). In contrast, the hysteroscopic morcellator system is larger (5.6mm outer diameter) and requires acquisition of specific hysteroscopes with an offset proximal eyepiece to allow the rigid mechanical cutting device to be inserted in direct alignment with the barrel of the hysteroscope. Thus in an outpatient setting, the bipolar electrode may have advantages over the larger hysteroscopic morcellator in terms of ease of uterine instrumentation.

In view of the development of hysteroscopic morcellation and potential advantages associated with this innovation in hysteroscopic instrumentation, the investigators believe that there is an urgent need to undertake a robust health technology assessment. It is timely to perform an RCT now before the findings of the OPT trial are available (which will recommend outpatient as opposed to day-case treatment if increased cost-effectiveness is demonstrated). If the morcellator is considered an easier technology to use by gynaecologists (i.e. less operator skill required), then there is a danger that it will become widely adopted for outpatient use without supporting evidence of benefit.

ELIGIBILITY:
Inclusion Criteria:

* Finding of a benign polyp on diagnostic hysteroscopy
* Patient considered able to tolerate outpatient hysteroscopic polypectomy based upon the response to preliminary diagnostic hysteroscopy. NB. all polyps diagnosed at hysteroscopy will be considered feasible to remove in the outpatient setting regardless of size, location or number. Patient factor(s) will be the only exclusion criteria following the diagnosis of benign, uterine polyp(s).
* Need for polypectomy
* Written informed consent

Exclusion Criteria:

• Hysteroscopic features suggesting malignant lesion

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The time taken for polyp removal | at the time of surgery (day 1 intraoperatively)
  The time taken to remove the polyp will be defined as the time from insertion to removal of vaginal instrumentation post-randomisation

SECONDARY OUTCOMES:
Patient acceptability or pain | immediately after the surgery (day 1)
  The acceptability of the trial will be assessed a questionnaire using pain visual analogue scores. The patient will be given a preoperative questionnarie to get a pain baseline and this will be followed postoperative pain questionnaire.
Completion of polyp removal | at the time of surgery (day 1 intraoperatively)
  A complete uterine polypectomy will be defined as the detachment and retrieval of all visible polyp tissue (single or multiple polyps), such that no polyp remnants remain within the uterine cavity. An incomplete procedure will include any of the following: (i) failure to detach any polyp tissue from the uterine wall; (ii) partial detachment of polyp(s) from the uterine wall and (iii) failure to retrieve the detached specimen from the uterine cavity

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Clark, MBChB, Principal Investigator — Birmingham Womens Hospital
Locations (1):
- Birmingham Womens Hospital, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Smith PP, Middleton LJ, Connor M, Clark TJ. Hysteroscopic morcellation compared with electrical resection of endometrial polyps: a randomized controlled trial. Obstet Gynecol. 2014 Apr;123(4):745-51. doi: 10.1097/AOG.0000000000000187. PMID 24785600